CLINICAL TRIAL: NCT02508987
Title: Obesity and Oxidative Stress in Patients With Different Periodontal Status: A Cross-sectional Study
Brief Title: Obesity and Oxidative Stress in Patients With Different Periodontal Status
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Vadim Ekrem Atabay, phd, Ondokuz Mayıs University
Other Study IDs: PYO.DIS.1904.13.002
Record Dates: First submitted 2015-07-22; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Obesity; Periodontitis; Gingivitis
Keywords: Obesity; oxidative stress; antioxidants; periodontal disease
MeSH Terms: conditions — Obesity; Periodontitis; Gingivitis; Periodontal Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — gingival crevicular fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Group 1: Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions as periodontally healthy.Periodontal status was determined by evaluating the following clinical parameters: Silness & Löe plaque index; Löe & Silness gingival index; probing pocket depth; clinical attachment level; bleeding on probing.
  Obesity was diagnosed according to World Health Organization criteria using body mass index. 18.50-24.99 kg/m2: Normal-weight
- Group 2: Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions as gingivitis. Periodontal status was determined by evaluating the following clinical parameters: Silness & Löe plaque index; Löe & Silness gingival index; probing pocket depth; clinical attachment level; bleeding on probing.
  Obesity was diagnosed according to World Health Organization criteria using body mass index.
  18.50-24.99 kg/m2: Normal-weight
- Group 3: Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions as 'generalized chronic periodontitis'. Periodontal status was determined by evaluating the following clinical parameters: Silness & Löe plaque index; Löe & Silness gingival index; probing pocket depth; clinical attachment level; bleeding on probing.
  Obesity was diagnosed according to World Health Organization criteria using body mass index.18.50-24.99 kg/m2: Normal-weight
- Group 4: Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions as either 'periodontally healthy'. Periodontal status was determined by evaluating the following clinical parameters: Silness & Löe plaque index; Löe & Silness gingival index; probing pocket depth; clinical attachment level; bleeding on probing.
  Obesity was diagnosed according to World Health Organization criteria using body mass index. 30.00-34.9 kg/m2: Obesity class I
- Group 5: Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions as 'gingivitis'. Periodontal status was determined by evaluating the following clinical parameters: Silness & Löe plaque index; Löe & Silness gingival index; probing pocket depth; clinical attachment level; bleeding on probing.
  Obesity was diagnosed according to World Health Organization criteria using body mass index. 30.00-34.9 kg/m2: Obesity class I
- Group 6: Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions as 'generalized chronic periodontitis'. Periodontal status was determined by evaluating the following clinical parameters: Silness & Löe plaque index; Löe & Silness gingival index; probing pocket depth; clinical attachment level; bleeding on probing.
  Obesity was diagnosed according to World Health Organization criteria using body mass index. 30.00-34.9 kg/m2: Obesity class I

SUMMARY:
The aim of the study is to evaluate the effect of obesity on periodontally healthy or diseased tissues.Normal weight and obese subjects were analyzed in 6 groups. Clinical periodontal status was determined through plaque index, gingival index, bleeding on probing, pocket probing depth, clinical attacment level and radiographs.

Oxidative stress is known to contribute to various diseases by affecting cellular functions through the oxidation of proteins, lipids and DNA. Oxidative stress can be assessed by measuring the products of oxidative damage found in proteins, lipids and DNA or reductions in total antioxidant capacity Malondialdehyde, protein carbonyl and total antioxidant capacity levels are biomarkers of oxidative stress in gingival crevicular fluid.

DETAILED DESCRIPTION:
This cross-sectional study was conducted with 93 subjects (45 normal-weight, and 48 class I obese) recruited from the Periodontology Department at the Ondokuz Mayıs University Faculty of Dentistry; Endocrinology and Metabolic Diseases Department at the Ondokuz Mayıs University Faculty of Medicine in Turkey, between September 2012 and March 2014.

The study protocol was approved by the Local Ethics Committee, and written informed consent was obtained from all study participants in accordance with the Helsinki Declaration (revised in 2000).

Oxidative stress occurs when the balance between reactive oxygen species and antioxidants become unbalanced. OS can be determined by evaluation of oxidative damage products in proteins, lipids and DNA or the reduction of total antioxidant capacity.

Malondialdehyde level is the biomarker of oxidative stress in lipids. Protein carbonyl level is the biomarker of oxidative stress in proteins.Total antioxidant capacity level is another biomarker of oxidative stress. Malondialdehyde, protein carbonyl and total antioxidant levels in crevicular fluid were examined by ELISA method.

Obesity was diagnosed according to World Health Organization criteria using body mass index. Body mass index is defined as a person's weight, in kilograms (kg), divided by the square of height in meters (m), and it is classified as follows:

≤18.49 kg/m2: Under-weight 18.50-24.99 kg/m2: Normal-weight 25.00-29.99 kg/m2: Overweight 30.00-34.9 kg/m2: Obesity class I 35.00-39.99 kg/m2: Obesity class II

≥40.00 kg/m2: Obesity class III (morbid obesity)

Periodontal status was determined through plaque index, gingival index, bleeding on probing, pocket probing depth, clinical attachment level and radiographs. Periodontal status was classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions as either 'periodontally healthy', 'gingivitis' or 'generalized chronic periodontitis'. Study participants were then grouped according to body mass index and periodontal status as follows:

Group 1: Group normal weight +periodontally healthy subjects Group 2: Group normal weight + gingivitis subjects Group 3: Group normal weight + generalized chronic periodontitis subjects Group 4: Group obese + periodontally healthy subjects Group 5: Group obese + gingivitis subjects Group 6: Group obese + generalized chronic periodontitis subjects All clinical examinations and gingival crevicular fluid collection were performed by a single examiner. All laboratory procedures were performed by another researcher blinded to the study.

A total of 108 gingival crevicular fluid samples were taken from the Group 5 (18 subjects x 6 sites) and 90 samples from each of the remaining 5 groups (15 subjects per group x 6 sites). All samples were collected between 8-10 am on the day following periodontal status assessment. Samples were collected from the sites in the chronic periodontitis group that fit the following criteria: pocket probing depth≥5mm, clinical attachment level≥5mm and ≥30% radiographic alveolar bone loss. Accordingly, gingival crevicular fluid samples were collected from 2 molar teeth, 2 premolar teeth and 2 incisors. Gingival crevicular fluid samples were collected from the same 6 sites in the gingivitis and periodontally healthy groups in order to maintain consistency of sampling.

ELIGIBILITY:
Inclusion Criteria:

(i) ≥ 18 years of age and having ≥ 16 teeth; (ii) no periodontal therapy in the 6 months prior to data collection; (iii) no systemic problems or chemotherapy within the 6 weeks prior to data collection; (iv) no previous history of smoking.

Exclusion Criteria:

(i) medical history of cancer, rheumatoid arthritis, diabetes mellitus, or cardiovascular disease; (ii) compromised immune system; (iii) pregnancy, menopause, or lactation; (iv) ongoing drug therapy that might affect the clinical characteristics of periodontitis; (v) use of systemic antimicrobials during the 6 weeks prior to data collection; (vi) dental treatment during the 6 months prior to data collection.

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Systemically healthy 45 normal weight adults and 48 class I obese adults
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde levels in gingival crevicular fluid as measured an oxidative stress marker in lipids | between 8-10 am on the day following periodontal status assessment.
  Malondialdehyde is the most specific and most used molecule for measurement of biological lipid oxidation.
Protein Carbonyl levels in gingival crevicular fluid as measured an oxidative stress marker in proteins | between 8-10 am on the day following periodontal status assessment.
  Protein carbonyl is another biomarker of oxidative stress
Reduction of total antioxidant capacity levels in gingival crevicular fluid as measured an oxidative stress marker | between 8-10 am on the day following periodontal status assessment.
  Total antioxidant capacity provides an overview of the biological interaction between an individuals' antioxidant status and how well these antioxidants are able to protect host cells during periods of oxidative stress. Due to the potential synergistic effects of different antioxidant molecules, the measurement of total antioxidant capacity can provide a more accurate assessment of antioxidant status than the separate measurement of individual molecules.

SECONDARY OUTCOMES:
Plaque index | the day before gingival crevicular fluid samples were collected
Gingival index | the day before gingival crevicular fluid samples were collected
Bleeding on probing | the day before gingival crevicular fluid samples were collected
Pocket probing depth | the day before gingival crevicular fluid samples were collected
Clinical attachment level | the day before gingival crevicular fluid samples were collected

CONTACTS AND LOCATIONS:
Overall Officials: Vadim E Atabay, phd, Principal Investigator — research assistant

REFERENCES:
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464